CLINICAL TRIAL: NCT02061202
Title: Inhaled Mometasone to Promote Reduction in Vasoocclusive Events
Brief Title: Inhaled Mometasone to Reduce Painful Episodes in Patients With Sickle Cell Disease
Acronym: IMPROVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey Glassberg (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey Glassberg, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 12-1565; K23HL119351 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-02-12 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Pain Crisis; Painful Crisis; Sickle Pain
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mometasone Furoate (Experimental): 1 puff daily (220mcg) for 16 weeks
  Interventions: Drug: Mometasone Furoate
- Placebo (Placebo Comparator): 1 puff daily for 16 weeks. Training inhaler that does not contain any medication (placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate — inhaled cortico-steroid (ICS) with a dosage of 220mcg once daily for 16 weeks
  Arms: Mometasone Furoate
Drug: Placebo — placebo training inhaler with the same instructions as the experimental group.
  Arms: Placebo

SUMMARY:
The proposed research is designed to test the global hypothesis that inhaled corticosteroids (ICS), a therapy developed to treat asthma, will prevent vasoocclusive painful episodes in adults with Sickle Cell Disease (SCD) who wheeze, but do not meet criteria for a diagnosis of asthma. The specific aims of this proposal are 1) Conduct a feasibility study - a randomized controlled trial of ICS for adults with SCD who do not meet criteria for a diagnosis of asthma but report recurrent cough or wheezing, 2) Measure the effects of ICS on biological correlates of pulmonary inflammation (as determined by exhaled nitric oxide) and vascular injury (as determined by sVCAM) in SCD, and 3) Compare properties of traditional and Bayesian adaptive clinical trial design for therapeutic trials in SCD in preparation for designing a definitive trial of ICS. These aims have the potential to 1) change the standard of care for individuals with SCD and recurrent cough or wheeze, 2) provide insight into the pathogenesis of non-asthmatic wheezing in SCD and its response to treatment, 3) explore the suitability of innovative clinical trial designs to overcome the challenges that have hindered therapeutic innovation for SCD.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 or older
* Sever SCD phenotypes (Hb SS and Sβthalassemia0)
* A positive response to cough/wheeze questions

Exclusion Criteria:

* Patient carries a physician diagnosis of asthma
* Patient is prescribed asthma medications
* Patient is currently having a painful crisis (as defined by validated pain diary questions)
* Patient has acute respiratory symptoms
* Known hypersensitivity to milk proteins
* Meets criteria for our operational diagnosis of asthma
* More than 15 ED visits for pain over the preceding 12 months
* Admitted or discharged from the hospital for SCD pain within the last 7 days

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Glassberg, MD, MA, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Langer AL, Leader A, Kim-Schulze S, Ginzburg Y, Merad M, Glassberg J. Inhaled steroids associated with decreased macrophage markers in nonasthmatic individuals with sickle cell disease in a randomized trial. Ann Hematol. 2019 Apr;98(4):841-849. doi: 10.1007/s00277-019-03635-9. Epub 2019 Feb 20. PMID 30783732
- [Derived] Glassberg J, Minnitti C, Cromwell C, Cytryn L, Kraus T, Skloot GS, Connor JT, Rahman AH, Meurer WJ. Inhaled steroids reduce pain and sVCAM levels in individuals with sickle cell disease: A triple-blind, randomized trial. Am J Hematol. 2017 Jul;92(7):622-631. doi: 10.1002/ajh.24742. Epub 2017 Jun 5. PMID 28370266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2014, with first enrollment in March 2014, and last enrollment in October 2016
Period: Overall Study
Arm/Group | Mometasone Furoate | Placebo
Started | 36 | 18
Completed | 35 | 17
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant in each group was lost to follow up prior to data collection and excluded from analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate | Placebo | Total
Number analyzed (Participants) | 35 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8.56) | 36 (9.81) | 32 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 6 | 24
  Male | 17 | 11 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Follow up
Description: Feasibility is determined by calculating the proportion of randomized participants who complete follow up and a minimum of 30 pain diaries with good adherence to the study medication vs. the number enrolled.
Time Frame: at 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 36 | 18
Participants | 35 | 17

2. Secondary Outcome: Change in Exhaled Nitric Oxide (eNO)
Description: Change in effects of inhaled corticosteroids (ICS) as measured by exhaled nitric oxide levels, which is the primary marker of pulmonary inflammation.
Time Frame: Before ICS therapy begins and at 8 weeks post enrollment
Measure: Mean (95% Confidence Interval); unit: ppb
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
ppb | 0.63 [-2.51 to 3.77] | 2.71 [0.48 to 5.90]

3. Secondary Outcome: Change in Soluble Vascular Cell Adhesion Molecule (sVCAM) Level
Description: Mean Change in effects of inhaled corticosteroids vascular injury, assessed by biomarker sVCAM as a surrogate for vascular injury.
Time Frame: Before ICS therapy begins and at 8 weeks post enrollment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
ng/mL | -182.47 (785.21) | 170.25 (182.39)

4. Secondary Outcome: Change in Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me)
Description: Mean changes in ASCQ-Me (NHLBI developed a patient-reported Sickle Cell Disease (SCD) quality of life measurement tool) pain impact, at week 20 as compared to baseline. A reduction change on a 100-point scale indicated improved quality of life. ASCQ-Me uses a T-score metric (0-100) in which 50 is the mean of the reference population and 10 is the standard deviation (SD) of that population.
Time Frame: baseline and week 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
score on a scale | 2.8 (22.7) | 6.9 (24.0)

5. Secondary Outcome: The Medication Adherence Report Scale
Description: The medication adherence report scale for asthma is a 10 question tool scored between 0 and 5, with full scale from 0 to 25, with higher scores indicating greater adherence
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
score on a scale | 17.7 (2.25) | 17.1 (1.78)

6. Secondary Outcome: Change in the Numerical Rating Scale (NRS) for Pain
Description: Mean change in patient reported pain NRS score, full scale range 0- 10, higher score indicate more pain
Time Frame: baseline and 20 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
score on a scale | 2.09 (2.55) | 2.82 (2.21)

7. Secondary Outcome: Asthma Control Test
Description: Asthma control test, total score from 0-25, with higher score indicating more symptoms
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
score on a scale | 17.7 (2.25) | 17.1 (1.78)

8. Secondary Outcome: Admissions or Visits to the Hospital
Description: Number of times participant visited the Emergency Department (ED) or was admitted to the hospital
Time Frame: baseline through 8 weeks
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
Events
  ED visits | 0.97 (1.52) | 1.12 (1.87)
  Observation admits | 0.37 (0.77) | 0.59 (1.18)
  Admissions | 0.37 (0.77) | 0.47 (1.23)

9. Secondary Outcome: Change in Reticulocytes Count
Description: Mean change in reticulocytes count - the number of new red blood cells.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: 10^3 cells/μL
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
10^3 cells/μL | -0.15 (0.39) | 0.07 (0.52)

10. Secondary Outcome: Change in FEV1/FVC
Description: Mean change in FEV1/FVC at 8 weeks compared to baseline
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mometasone Furoate | Placebo
Number analyzed (Participants) | 35 | 17
ratio | -0.71 (3.42) | -1.41 (3.39)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Mometasone Furoate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/17
Other Adverse Events (participants affected / at risk) | 15/35 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mometasone Furoate (N=35) | Placebo (N=17)
Hoarseness of voice (Respiratory, thoracic and mediastinal disorders) | 15 | 4
Thrush (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 15 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT02061202/Prot_SAP_000.pdf